CLINICAL TRIAL: NCT05478408
Title: Correlation of Mukbang Video Watching Behavior,Internet Addition and Mental Health Among General Population
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Wei XIA, PhD, Associate Professor, Sun Yat-sen University
Other Study IDs: L2022SYSU-HL-028
Record Dates: First submitted 2022-07-27; First posted 2022-07-28 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Mukbang
Keywords: Mukbang; Mental Health; Internet Addiction
MeSH Terms: conditions — Psychological Well-Being; Internet Addiction Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Questionnaires assessed general population: ① Internet users over the age of 18；
  ② Be able to read and communicate in Chinese.
  Interventions: Other: Questionnaires set

INTERVENTIONS:
Other: Questionnaires set — Participants will be asked to respond to the demographic information，the Depression Anxiety Stress Scale（DASS-21）and the Internet Addiction Test（IAT）.

SUMMARY:
This study will describe the general population's current situation of watching "Mukbang" videos, their mental health status and the level of Internet addiction tendency by means of an online survey, and analyze their correlations. It provides a theoretical basis for promoting healthy psychological development and standardizing management of "Mukbang" videos.

DETAILED DESCRIPTION:
Mental health issues have always been the focus of health management. The Lancet Global Commission on Mental Health and Sustainable Development also recommends a broad cross-sectoral approach to mental health issues. With the rapid development of short videos and self-media, watching "Mukbang" is a behavioral way for netizens to alleviate mental health problems such as anxiety and depression. However, watching "Mukbang" can be Internet addictive. At present, there is no research to predict the addictive behavior caused by "Mukbang", and there is no relevant research to explore its addiction mechanism. Although it has been clear that Internet addiction and mental health disorders are significantly related, there is no clear statement on whether there is a common risk factor, a mediating effect, or a causal relationship between the two. The behavior of watching "Mukbang" videos may be in a mediating position between the two. This study will further explore the relationship between the three based on the use and satisfaction theory.

ELIGIBILITY:
Inclusion Criteria:

* Internet users over the age of 18;
* Be able to read and communicate in Chinese.

Exclusion Criteria:

* Those who can not complete communication due to serious mental or physical diseases such as deafness, unclear consciousness caused by mental illness, etc.;

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: General Population
Sampling Method: Probability Sample
Enrollment: 2918 (Estimated)
Dates: Start 2022-08-15 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Features of Watching "Mukbang" Videos | Baseline
  The"Mukbang" watching features will be assessed by a questionnaire designed by the researcher and recorded by the subjects themselves, including watching time, watching rate, watching preferences and watching experience.
Mental Health | Baseline
  The mental health status will be assessed by the Depression Anxiety Stress Scale（DASS-21），4-point Likert rating scale, which contains 21 items to describe personal recent negative emotional experience. The full scale consists of three subscales of depression, anxiety and stress, each of which contains 7 items.
Internet Addiction | Baseline
  The Internet addiction risk will be assessed by the Chinese version of Young's self-rating Internet addiction scale，a total of 20 items. Each item used a 5-point Likert scale(1=rarely, 2=occasionally, 3=sometimes, 5=always), and the total score ranged from 20 to 100. The higher the score, the more serious the risk of Internet addiction.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Xia, PhD, Principal Investigator — Sun Yat-sen University
Locations (1):
- XIAW, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No